CLINICAL TRIAL: NCT00943553
Title: A Randomized Study of Epigenetic Priming Using Decitabine With Front Line Induction Chemotherapy Compared With Immediate Induction Chemotherapy in Pediatric Acute Myelogenous Leukemia (AML) Subjects.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by Sponsor
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7373-G000-201
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Acute Myelogenous Leukemia (AML)
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Induction Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: decitabine Induction Chemotherapy
- 2 (Experimental)
  Interventions: Drug: Induction Chemotherapy

INTERVENTIONS:
Drug: decitabine Induction Chemotherapy — Arm A - 12 days (5 days of intravenous (IV) decitabine 20 mg/m^2 followed by 7 days of induction chemotherapy with IV daunorubicin 45 mg/m^2 and cytarabine 100 mg/m^2/day)
  Other Names: E7373
  Arms: 1
Drug: Induction Chemotherapy — Arm B - 7 days (7 days of induction chemotherapy with IV daunorubicin 45 mg/m^2 and cytarabine 100 mg/m^2/day only)
  Other Names: E7373
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of decitabine when used before chemotherapy to treat leukemia in pediatric patients. The study will also evaluate the ways decitabine is affected or changed when used in the human body.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age 1 to16 years, inclusive
2. Females of childbearing potential must have a negative serum beta human chorionic gonadotropin (β-hCG) at Visit 1 (Screening) and a negative urine pregnancy test prior to starting study drugs (Visit 2). Female subjects of childbearing potential must agree to be abstinent or to use a highly effective method of contraception (eg, condom + spermicide, condom + diaphragm with spermicide, intrauterine devise (IUD), or have a vasectomised partner) for at least one menstrual cycle prior to starting study drug(s) and throughout the longer of either Core Study period or 30 days after the last dose of study drug. Those females using hormonal contraceptives must also be using an additional approved method of contraception (as described previously).
3. Sexually mature male patients who are not abstinent or have not undergone a successful vasectomy, who are partners of women of childbearing potential must use, or their partners must use a highly effective method of contraception (eg, condom + spermicide, condom + diaphragm with spermicide, IUD) starting for at least one menstrual cycle prior to starting study drug(s) and throughout the entire study period and for 30 days (longer if appropriate) after the last dose of study drug. Those with partners using hormonal contraceptives must also be using an additional approved method of contraception (as described previously).
4. Diagnosis of acute myelogenous leukemia (AML)(bone marrow or peripheral blood blasts ≥ 20%)
5. Adequate cardiac function as defined by an echocardiogram or multiple gated acquisition (MUGA) scan demonstrating an ejection fraction within normal limits
6. Are willing and able to comply with all aspects of the protocol
7. Provide written informed consent from subject's guardian or legally authorized representative and child assent (if applicable)

Exclusion Criteria:

1. Females who are pregnant (positive β-hCG test) or lactating
2. History of chronic myelogenous leukemia (CML) [t(9;22)]
3. Acute promyelocytic leukemia (M3 subtype in French-American-British [FAB] classification).
4. Known central nervous system (CNS) leukemia
5. AML associated with congenital syndromes such as Down syndrome, Fanconi anemia, Bloom syndrome, Kostmann syndrome, or Diamond Blackfan anemia
6. White blood cell (WBC) count > 40,000/mm3
7. Serum creatinine > 2.5 mg/dL
8. Alanine aminotransferase (ALT) > 5 x upper limit of normal (ULN) and/or total bilirubin > 3 x ULN
9. Prior chemotherapy (other than hydroxyurea) or radiation therapy for AML
10. Known to be human immunodeficiency virus (HIV) positive
11. Any history of or concomitant medical condition that, in the opinion of the Investigator, would compromise the subject's ability to safely complete the study
12. The Investigator believes the subject to be medically unfit to receive the study drug or unsuitable for any other reason.
13. Subject with hypersensitivity to decitabine, daunorubicin, or cytarabine
14. Has participated in a drug trial in the last 4 weeks

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint (Core Component): Complete Remission (CR) Rate as defined by International Working Group - 2003 criteria | ~ 2 years

SECONDARY OUTCOMES:
Secondary Endpoint (Core Component): Methylation of DNA following decitabine therapy. | Until Week 3 after chemotherapy
Secondary Endpoint (Core Component): Time to platelet recovery (≥ 100,000/mm3) and time to neutrophil recovery (absolute neutrophil count [ANC] ≥ 1000/mm3) following induction chemotherapy | Until ~ 4 weeks after last dose of induction chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Peter Tarassoff, MD, Study Director — Eisai Inc.
Locations (1):
- New Delhi, New Delhi, India